CLINICAL TRIAL: NCT04637659
Title: E. Faecalis Prevalence in Primary and Secondary Endodontic Infections: a Pre-post Microbial Analysis Following Chemo-mechanical Preparation
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Professor, University of Siena
Other Study IDs: EF001
Record Dates: First submitted 2020-11-13; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — For each patient 4 samples will be taken with sterile paper cones: saliva sample before the endodontic treatment, canal sample pre and post treatment, negative control in the rubber dam.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy non-treated teeth: Healthy teeth being treated for restorative or prosthodontics reasons
  Interventions: Procedure: Root Canal Treatment
- Healthy treated teeth: Teeth being retreated for restorative or prosthodontics reasons
  Interventions: Procedure: Root Canal Treatment
- Irreversible pulpitis: Teeth being treated because of a poor pulpal status
  Interventions: Procedure: Root Canal Treatment
- Post-treatment apical periodontitis: Teeth being retreated due to the presence of an apical lesion
  Interventions: Procedure: Root Canal Treatment
- Necrosis: Teeth being treated because of pulpal necrosis
  Interventions: Procedure: Root Canal Treatment

INTERVENTIONS:
Procedure: Root Canal Treatment — Chemo-mechanical preparation will be performed using reciprocating instruments . Irrigation will be carried out with 5.25% NaOCl during instrumentation and a final flush of 17% EDTA followed by 5.25% NaOCl. After drying with paper points, canal obturation will be achieved through continuous condensation wave technique. Obturation with gutta-percha will be performed using Reciproc blue R25 master cones and root canal sealer using the BeeFill 2 in 1 device (VDW, GmbH) with a small heat carrier (#40 tip size and .03 taper) following the manufacturer's instructions. After the down-packing phase, the back-filling will be performed with the same device and manual compaction using endodontic pluggers.

SUMMARY:
Post-treatment apical periodontitis is a fairly prevalent condition frequently caused by a persistent endodontic infection due to failure of the endodontic treatment. Microbial species in treated or untreated root canals were found to be different, with the former being less diverse and mainly characterized by Gram positive, facultative anaerobes bacteria than the latter. Enterococcus faecalis is the most frequently detected species in root-filled teeth in many studies (Zhang et al., 2015). In fact, E. Faecalis retains many virulence factors allowing adhesion to host cells and extracellular matrix, tissue invasion and damage through toxins release, as well as the ability to survive even in harsh environmental conditions. Further studies are needed to clarify E. faecalis prevalence among the different forms of pulpal and periapical lesions as well as its correlation with clinical symptoms.

ELIGIBILITY:
Inclusion criteria:

* between the ages of 18 and 70;
* good systemic health.
* patients in need of an endodontic treatment/retreatment

Exclusion criteria:

* taking antibiotic therapy in the previous 3 months;
* presence of communication between the canal system and the oral cavity;
* teeth that are not perfectly isolated;
* teeth with probing depth >4 mm with positive BOP.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients in need of an endodontic treatment and meeting the inclusion/exclusion criteria will be eligible for the inclusion in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of E.Faecalis in the canal before the treatment for each group | Pre-treatment microbial sampling in the canal was carried out 1 day once arrived at working length with a 10 K-file
  E.Faecalis prevalence in the canal before the treatment will be calculated for each group.

SECONDARY OUTCOMES:
Correlation between E.Faecalis presence in the canal before the treatment and the pulpal/periapical status | Pre-treatment microbial sampling in the canal was carried out 1 day once arrived at working length with a 10 K-file
  Correlation between E. faecalis presence in the canal before the treatment and the pulpal/periapical status for each group will be calculated through measures of association

OTHER OUTCOMES:
Correlation between E. Faecalis presence in the canal before the treatment and its presence in saliva (pre-treatment) | Pre-treatment microbial sampling in saliva was carried out 1 day before rubber dam isolation. Pre-treatment microbial sampling in the canal was carried out once arrived at working length with a 10 K-file.
  Correlation between E. Faecalis presence in the canal before the treatment and its presence in saliva (pre-treatment) will be calculated
Ability of the endodontic treatment to remove E. Faecalis from the canal | Pre-treatment microbial sampling in the canal was carried out 1 day once arrived at working length with a 10 K-file. Post treatment microbial sampling will be carried out at the end of the endodontic treatment after the final wash with EDTA and NaOCl
  Pre-post endodontic treatment comparison as to E. Faecalis presence in the canal will be carried out
Correlation between the presence of E. Faecalis in the canal before the treatment and the presence of a radiographic lesion | Pre-treatment microbial sampling in the canal was carried out 1 day once arrived at working length with a 10 K-file
  Correlation between the presence of E. Faecalis in the canal before the treatment and the presence of a radiographic lesion (measured with the PAI score)

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, Italy

IPD SHARING:
Plan to Share IPD: Undecided